CLINICAL TRIAL: NCT06309576
Title: Experimental Approach to Test Predictions of Body Weight Regulation Models
Acronym: DIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Tulane University (Other)
Responsible Party: Principal Investigator, Rodrigo Fernandez-Verdejo, Visiting Assistant Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 2023-069
Record Dates: First submitted 2024-03-01; First posted 2024-03-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Underweight
Keywords: Energy expenditure; Energy intake; Energy balance; Set point model; Dual-intervention point model
MeSH Terms: conditions — Obesity; Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting-refeeding cycle (Experimental): Participants will be maintained in metabolic chambers and exposed to 1 day of energy balance, 2 days of fasting, and 2 days of ad-libitum refeeding.
  Interventions: Behavioral: Fasting-refeeding cycle

INTERVENTIONS:
Behavioral: Fasting-refeeding cycle — Participants will be maintained in metabolic chambers and exposed to 1 day of energy balance with a standard diet, 2 days of fasting (only water), and 2 days of ad-libitum refeeding using a liquid diet provided in hydration bladders to avoid portion control.

SUMMARY:
The regulation of human body weight and fatness is not fully understood. Although some models of regulation have been proposed (set point, dual-intervention point, others), no studies have been designed to test their predictions. In this pilot and feasibility study, the investigators will implement an experimental approach to test the predictions of models of body weight regulation in humans. Men and women with either low body weight or obesity will be exposed to a 2-day fasting followed by a 2-day ad-libitum refeeding. During the entire fasting-refeeding period, energy intake and expenditure will be accurately measured within metabolic chambers. The investigators will therefore determine the compensatory responses to fasting elicited to prevent weight loss. The results will serve to design and power future studies to better understand body weight regulation.

DETAILED DESCRIPTION:
Background:

Although body weight regulation models have been proposed, experimental approaches for testing their predictions are lacking. The set point (SP) model proposes that a biologically determined fatness is defended by activating compensatory responses to prevent its change. The dual-intervention point (DIP) model proposes that there are two levels of fatness (lower and upper intervention points) within which fatness is weakly regulated. Compensatory responses would only be activated once the lower or upper intervention points are reached. In response to prolonged fasting, the SP model predicts the compensatory responses to be independent of the initial body weight. In contrast, the DIP model predicts higher responses in individuals who are closer to the lower intervention point (low body weight) compared to those who are farther away (obesity). None of these models predicts a different response in men vs. women. Our pilot and feasibility study will implement an experimental approach to test these predictions in humans by thoroughly measuring compensatory responses in energy expenditure and energy intake.

Design:

Twelve individuals (3 men with low body weight and 3 with obesity; 3 women with low body weight and 3 with obesity) will be kept inpatient in metabolic chambers for 5 consecutive days and exposed to a 1-day energy balance, 2-day fasting, and 2-day ad-libitum refeeding. The primary outcome will be the extent of compensatory response, calculated as the cumulative energy balance during the 5-day inpatient period.

Objectives:

1. To determine the extent of compensatory response induced by a 2-day fasting followed by a 2-day ad-libitum refeeding in humans overall and among different subgroups (low body weight, obesity, men, women).
2. To explore the timing of the compensatory responses during a 2-day fasting followed by a 2-day ad-libitum refeeding in humans.
3. To explore potential physiological determinants of the inter-individual variability in the compensatory response induced by a 2-day fasting followed by a 2-day ad-libitum refeeding in humans.

Relevance:

Understanding how body weight is regulated in humans can help to prevent or treat obesity. In this pilot and feasibility study, the investigators propose an experimental approach to test the predictions of two body weight regulation models in response to fasting and explore potential sex differences. These preliminary data will be used to design and power future studies for testing models of body weight regulation in humans.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index lower than 20 kg/m2 for the low body weight group, or 30 kg/m2 or greater for the obesity group
* 18-40 years old
* Nulliparous and regular menstrual cycle (25-35 days) during the last six months (in women)
* Normal thyroid function, blood count, and chemistry 15 panel (normal plasma glucose will be considered at <100 mg/dL; normal serum HDL cholesterol at >=50 mg/dL for women and >=40 mg/dL for men; and normal serum triglycerides at <150 mg/dL).
* Self-reported weight stability during the last six months (±3 kg)
* Rate the liking of at least one of the flavored liquid meals (Ensure Plus, Abbot Nutrition) between 5 and 8 on a 9-point Likert scale
* Willing to only drink up to two assigned flavors of Ensure Plus for two consecutive days

Exclusion Criteria:

* Eating disorders as indicated by a global score ≥2.80 in the Eating Disorder Examination Questionnaire, or a previous diagnosis of an eating disorder
* For the low body weight group, having food insecurity (with or without hunger) as assessed by the USDA
* Recreational moderate-intensity physical activity ≥150 min/week, recreational vigorous-intensity physical activity ≥75 min/week, or a combination of recreational moderate-intensity and vigorous-intensity physical activity (moderate time + [2 × vigorous time]) ≥150 min/week as assessed by the Global Physical Activity Questionnaire, or being a professional athlete
* Cigarette or vape smoking
* Intake of more than 14 alcoholic drinks per week
* Use of medications that may affect energy intake and/or expenditure, for example, semaglutide, liraglutide, exenatide, other GLP-1 receptor agonists, phentermine-topiramate, naltrexone-bupropion, orlistat, metformin, SGLT2 inhibitors, pramlintide, levocarnitine, amphetamines, and amphetamine-like drugs
* Human immunodeficiency virus, galactosemia, and lactose intolerance
* Diseases that affect energy homeostasis including endocrine such as hypo/hyperthyroidism, or type 1 or 2 diabetes; cancer; chronic pulmonary diseases; cardiovascular disease; and renal disease
* History of inflammatory bowel disease (ulcerative colitis, Crohn's), malabsorption syndromes (intestinal, pancreatic), and sprue or gluten intolerance
* Having moderate to severe sleep apnea defined as an oxygen desaturation index >10 times/hour assessed by overnight oximetry to be conducted on the night following the screening visit
* Use of oral hormonal contraceptives or less than 6 months using a hormonal intrauterine device (in women)
* Adults who are unable to consent
* Prisoners
* Currently pregnant or breastfeeding (in women)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Compensatory response | The cumulative energy balance is calculated one time using the data of 5 inpatient days
  Cumulative energy balance during the fasting-refeeding cycle

SECONDARY OUTCOMES:
Timing of the compensatory response | The cumulative energy balance calculated for the following time periods along the 5-day fasting-refeeding cycle: day 1 to 2, day 1 to 3, day 1 to 4, during fasting (day 2 to 3), and during refeeding (day 4 to 5)
  Cumulative energy balance during different time periods of the 5-day fasting-refeeding cycle
Protein balance | Protein balance is calculated one time using the data of 5 inpatient days
  Protein balance (intake minus oxidation) during the fasting-refeeding cycle
Carbohydrate balance | Carbohydrate balance is calculated one time using the data of 5 inpatient days
  Carbohydrate balance (intake minus oxidation) during the fasting-refeeding cycle
Lipid balance | Lipid balance is calculated one time using the data of 5 inpatient days
  Lipid balance (intake minus oxidation) during the fasting-refeeding cycle
Overall appetite | Overall appetite is measured 8 times per day (every 2 hours from approximately 8:00 AM) during the 5 inpatient days
  Calculated from the results of visual analog scales that record hunger, satiety, fullness, and prospective food consumption
Food preference | Measured once a day, in the fasting state (at approximately 8:00 AM), during the 5 inpatient days
  Measured using the Food Preference Questionnaire
Physical activity | Measured continuously (i.e. for 24 hours) every day during the 5 inpatient days
  Measured with wrist-worn accelerometers
Sleeping metabolic rate | Measured every day during the 5 inpatient days
  Measured within the metabolic chamber, between 2:00 and 5:00 AM, and extrapolated to 24 hours
Leptin | Measured once a day, in the fasting state (at approximately 8:00 AM), during the 5 inpatient days
  Circulating concentrations of leptin
Appetite-regulating hormones | Measured once a day, in the fasting state (at approximately 8:00 AM), during the 5 inpatient days
  Circulating concentrations of ghrelin and insulin
Metabolites | Measured once a day, in the fasting state (at approximately 8:00 AM), during the 5 inpatient days
  Circulating concentrations of glucose, fatty acids, ketone bodies
Thyroid axis | Measured once a day, in the fasting state (at approximately 8:00 AM), during the 5 inpatient days
  Circulating concentrations of T4

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Fernandez-Verdejo, PhD, Principal Investigator — Pennington Biomedical Research Center; Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center; Dragana Lovre, MD, Principal Investigator — Tulane University
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected will be shared upon appropriate request as part of the NORC repository of Pennington Biomedical Research Center
Supporting Information: Study Protocol, ICF
Time Frame: After publication of the results for the main outcome
Access Criteria: Upon appropriate request
URL: https://my.pbrc.edu/NORC/NORCRepository/Landing/